CLINICAL TRIAL: NCT05497180
Title: Use of Passive Myofunctional Appliances for Snoring and Mild Obstructive Sleep Apnea
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 00117371
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Mandibular Advancement Devices; Myofunctional Therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Passive Myofunctional Appliance (Experimental): provision of passive myofunctional appliance
  Interventions: Device: passive myofunctional appliance
- Oral Appliance Therapy (Active Comparator): provision of mandibular advancement device
  Interventions: Device: standard oral appliance

INTERVENTIONS:
Device: passive myofunctional appliance — passive myofunctional appliance
  Arms: Passive Myofunctional Appliance
Device: standard oral appliance — standard oral appliance
  Arms: Oral Appliance Therapy

SUMMARY:
It is unknown whether passive myofunctional appliances can be used for the treatment of obstructive sleep apnea and snoring, nor how to select the appropriate size per individual patient. Exploring the possibility of using passive myofunctional appliances as a treatment option for patients with mild obstructive sleep apnea and/or snoring should be considered, especially as the time to fabricate and deliver custom designed dental sleep appliances can be significant (sometimes over a month). Use of passive myofunctional appliances as a transitional appliance or potentially as direct treatment for obstructive sleep apnea may significantly decrease time to treatment and also provide a less expensive treatment option for patients with obstructive sleep apnea. The purpose of this study is to determine whether passive myofunctional appliances can be used as a treatment option for patients suffering from snoring and mild obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
Obstructive sleep apnea is a medical condition where a person has great difficulty with breathing, or stops breathing all together, while asleep. This is a medical condition for which one of the current standard treatments is the use of a custom made dental appliance to help hold the person's airway open while asleep so that the person does not suffocate while sleeping. Current methodology within dentistry is to position the mandible somewhere approximately 70% of the person's maximum ability to position their mandible forward as the starting point (George Gauge technique), and then slowly move the bottom jaw forward as necessary. Recent literature (including that published by our team) has shown that different mandibular positioning techniques may require less protrusion, less titrations, and potentially decreased side effects compared with the traditional protrusive techniques. One of the most promising techniques involves the use of speech to determine mandibular position. The sibilant phenome technique would not require that a patient place their jaw outside of their normal functional range, and could potentially decrease the face pain/jaw joint problems commonly associated with the use of oral sleep appliances for the treatment of obstructive sleep apnea.

Myofunctional therapy has been shown to be effective at reducing sleep apnea disease indices for patients with obstructive sleep apnea. It can be thought of as targeted physiotherapy for the face, neck, and mouth muscles (including the lips, cheeks, and tongue). Due to its effectiveness and ability to reduce sleep apnea disease indices by up to 50%, it is considered an effective adjunctive treatment for obstructive sleep apnea. Recently, appliances made to aid in tongue, cheek, lip, and jaw positioning for myofunctional therapy have come onto the market. These are known as passive myofunctional appliances, and are prefabricated with varying sizes available.

It is unknown whether passive myofunctional appliances can be used for the treatment of obstructive sleep apnea and snoring, nor how to select the appropriate size per individual patient. Exploring the possibility of using passive myofunctional appliances as a treatment option for patients with mild obstructive sleep apnea and/or snoring should be considered, especially as the time to fabricate and deliver custom designed dental sleep appliances can be significant (sometimes over a month). Use of passive myofunctional appliances as a transitional appliance or potentially as direct treatment for obstructive sleep apnea may significantly decrease time to treatment and also provide a less expensive treatment option for patients with obstructive sleep apnea. The use of the sibilant phoneme technique may be used for determining the appropriate sizing for which passive myofunctional appliances may be appropriate for individual patients, or if no appropriate sizes are available for use.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with mild obstructive sleep apnea or snoring without sleep apnea.
* Patients 18 years or older
* Patients able to provide consent to treatment and participation in the study

Exclusion Criteria:

* Patients previously diagnosed as non-responders to oral appliance therapy for their sleep apnea
* Patients undergoing other active therapies for their sleep apnea
* Patients with a history of airway/sleep breathing surgical interventions
* Participants with a history of airway/sleep breathing surgical intervention are not eligible to be a part of this study do to risk of skewing test results
* Patients with craniofacial, syndromic, or neuromuscular disorders
* Patients with acute medical conditions requiring immediate attention
* Participants with an acute medical problem will be immediately referred to an appropriate physician and will not be allowed to enroll in the study until their health conditions are stable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-07-23 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Snoring volume | 3 months
  Decibel volumetric recordings with SnoreLab app

CONTACTS AND LOCATIONS:
Locations (1):
- Enjoy Dental, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No